CLINICAL TRIAL: NCT05825716
Title: Ifaa Effectiveness Evaluation: A Comparison of Multisectoral Food Security and Resilience Interventions in the Oromia Region of Ethiopia
Brief Title: Ifaa Effectiveness Evaluation on Food Security and Nutrition
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: IRB00023765
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Nutritional Wasting; Nutritional Stunting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ifaa Basic: comparison group
  Interventions: Other: Ifaa Basic
- Ifaa Enhanced: intervention group 1
  Interventions: Behavioral: Ifaa Enhanced
- Ifaa Enhanced + Livelihoods: intervention group 2
  Interventions: Other: Ifaa Enhanced + Livelihoods

INTERVENTIONS:
Other: Ifaa Basic — * PSNP Systems: (1) Provision of food aid commodities (wheat, oil, and pulse) per the PSNP transfer schedule for 3-6 months; 2) Food System Taskforce (FSTF) capacity building, and 3) private sector engagement
  * Health and Nutrition: 1) Government of Ethiopia (GoE) basic health extension program; 2) GoE supportive supervision coaching; 3) GoE-led community social behavior change (SBC) sessions; and 4) Community Management of Acute Malnutrition (CMAM) Programming.
  * Water and Sanitation: 1) Water infrastructure development; 2) improved governance via water, sanitation and hygiene (WASH) committees; and 3) water source monitoring.
  * Natural Resource Management: 1) Public works projects; 2) community training in planning and sustaining community assets; 3) Implementation of the environment and social management framework; 4) enhance participation of watershed committees
  Groups: Ifaa Basic
Behavioral: Ifaa Enhanced — * PSNP Systems: 1) establishment and training of Community Technical Coordinating Forum; 2) Case management capacity building; and 3) private sector construction of infrastructure
  * Health and Nutrition:1) the Care Group Model approach; 2) home garden promotion; 3) the nutrition budget calculator; and 4) labor and time-saving technologies.
  * Community-level interventions are 1) adolescent nutrition school clubs; 2) religious leader mobilization and training vulnerable groups; 3) audio toolkit against harmful traditional practice; 4) enhanced SBC tools for health/nutrition promotion; 5) additional health extension programs
  * Water and Sanitation: 1) Community Led Total Sanitation and Hygiene; 2) WASH systems assessments and strengthening; 3) Ensuring water quality and safety via routine monitoring; 4) Private sector engagement of WASH-related businesses;
  Groups: Ifaa Enhanced
Other: Ifaa Enhanced + Livelihoods — * Additional resources provided to the groups, including 1) Engagement of Private Service Providers to enable access to sustainable credit and larger loans; 2) Financial Education using an expanded 'Smart Skills' curriculum focusing on savings, smart borrowing and effective financial management; and 3) Life Skills Training for Youth.
  * Additional supports include: 1) Seven Steps of Marketing Training; 2) Climate Smart Agriculture to reduce water needs and increase soil health and vegetation coverage; 3) Producers Groups and linkages to markets/suppliers/buyers; Selected financial institutions will be provided with a credit guarantee fund and capacity-building support to help facilitate loans. Private sector value chain assessment and financing. Additional private sector engagement and linkage facilitation.
  Groups: Ifaa Enhanced + Livelihoods

SUMMARY:
The Ifaa Project is a USAID-funded Resilience and Food Security Activity (RFSA) that is being implemented by Catholic Relief Services (CRS) and partners in the East Hararghe Zone of the Oromia Region in Ethiopia. Ifaa targets households that are participating in the Productive Safety Net Programme (PSNP) which is a social protection program administered by the Government of Ethiopia that provides food and cash assistance to vulnerable households. The Ifaa Project will deliver multi-sectoral programming in 241 kebeles (sub-districts) in nine woredas (districts) of East Hararghe Zone, however, intervention packages vary by location. The proposed effectiveness evaluation will quantify the impacts of three different intervention packages in terms of key project indicators in the areas of household food security, diet, and child nutrition.

DETAILED DESCRIPTION:
The Ifaa Project will deliver multi-sectoral programming in 241 kebeles (sub-districts) in nine woredas (districts) of East Hararghe Zone, however, intervention packages vary by location. The three Ifaa intervention packages that will be delivered to PSNP beneficiaries based on the beneficiaries residence location include: 1) the Ifaa basic package; 2) enhanced package without livelihoods; and 3) enhanced package with livelihoods. The proposed effectiveness evaluation will quantify the impacts of three different intervention packages in terms of key project indicators in the areas of household food security, diet, and child nutrition. As the Ifaa consortium learning partner, Johns Hopkins School of Public Health (JHSPH) has been requested to design an effectiveness evaluation of the different intervention packages to compare their outcomes among beneficiary households.

To align the evaluation with project aims, key project indicators are used as study outcome measures. The specific objectives of the evaluation are to quantify the impact of Ifaa interventions as follows:

1. At the household level, Poor or Borderline Food Consumption Score (FCS)
2. at the individual level, change in minimum dietary diversity among children <5 years A secondary objective is to examine Ifaa impacts on child nutrition indicators, including measures of both acute and chronic malnutrition.

A longitudinal cohort design will be used to compare the effectiveness of three Ifaa intervention packages among PSNP beneficiaries in Eastern Hararghe: 1) the Ifaa basic package; 2) enhanced package without livelihoods; and 3) enhanced package with livelihoods. Under this approach, the enrolled households will have either a pregnant woman or children <24 months of age. Households will be followed over a two-year period, with the baseline and endline survey conducted at a similar time in the calendar year to avoid seasonal changes in food security. The magnitude of change in key indicators over time will be assessed for each group; if needed, adjusted models will be used to account for baseline differences between groups.

ELIGIBILITY:
Inclusion Criteria:

* Households are PSNP clients
* Households are Ifaa Project beneficiaries that are planned participants in: 1) Savings and Internal Lending Communities (SILC) groups (Ifaa Basic); 2) SILC Groups AND Care Groups (Ifaa and Enhanced); or 3) SILC groups AND Care Groups AND a Livelihoods Pathway.
* Households have a pregnant woman OR at least one child <36 months of age
* Households have an adult member that is capable of giving informed consent and completing an interview

Exclusion Criteria:

* Child-headed households (all members age 17yrs or less)
* Individuals not mentally able to give informed consent and complete an interview

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The overall goal of the Ifaa Project is to improve food security of vulnerable households in targeted PSNP communities, contributing to a sustained reduction in rural poverty. To achieve this goal, Ifaa will provide additional multi-sectoral interventions to benefit further 60,000 PSNP households in the Oromia region, which is Ethiopia's largest, most populous region and also one of its poorest. The study population is PSNP beneficiaries that are participating in the Ifaa Project.
Sampling Method: Non-Probability Sample
Enrollment: 3317 (Actual)
Dates: Start 2023-05-21 (Actual); Primary Completion 2025-07-05 (Actual); Study Completion 2025-07-05 (Actual)

PRIMARY OUTCOMES:
Change in Poor or Borderline Food Consumption Score (%) | baseline, 2 years
  The food consumption score (FCS) reflects the diversity and frequency of household food and nutritional intake consumed in the seven days preceding the survey and is an indicator used globally. The consumption frequency of eight food groups is assessed in the preceding 7 days, and weighted scores for each food group are summed to calculate the FCS; a higher FCS score indicates better food security. Household food security status is categorized using the following thresholds: 0-28 poor; 28.5-42 borderline; and >42 for acceptable.
Change in minimum dietary diversity (%) | baseline, 2 years
  The minimum dietary diversity (MDD) score is a population-level indicator to assess diet diversity as part of infant and young child feeding (IYCF) practices. Data are gathered from a questionnaire administered to the child's caregiver, usually as part of the IYCF module. Respondents are asked to indicate whether or not the child consumed any food over the previous 24 hours from each of eight food groups. The seven food groups included in the questionnaire are: grains, legumes and nuts, dairy products, flesh foods, eggs, vitamin A rich fruits and vegetables, other fruits and vegetables.

SECONDARY OUTCOMES:
Change in the prevalence of stunting (%) | baseline, 2 years
  Children will be measured for length (cm) among children 6 to 23 months of age. The length measures will be used to create indices of length-for-age (LAZ) z-score based on the World Health Organization (WHO) child growth standard. The prevalence of stunting (%) is defined as LAZ<-2.
  The prevalence of stunting (%) among children in the Ifaa enhanced intervention, Ifaa enhanced + livelihoods intervention versus. Ifaa basic group at endline (2 year) adjusting for the difference in the prevalence of stunting (%) at baseline between two areas.
Change in the prevalence of wasting (%) | baseline, 2 years
  Children will be measured for length (cm) and weight (kg) among children months. The length and weight measures will be used to create indices of weight-for-length (WLZ) z-score based on the WHO child growth standards.
  The prevalence of wasting (%) among children in the Ifaa enhanced intervention, Ifaa enhanced + livelihoods intervention versus. Ifaa basic group at endline (2 year) adjusting for the difference in the prevalence of stunting (%) at baseline between two areas.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Doocy, PhD, Principal Investigator — Bloomberg School of Public Health, Johns Hopkins University, Baltimore, MD, USA, 21205
Locations (1):
- Seifu Tadesse, Addis Ababa, Ethiopia

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT05825716/Prot_SAP_000.pdf